CLINICAL TRIAL: NCT06914206
Title: Esketamine Intravenous Infusion Combined With Pulsed Radiofrequency of Dorsal Root Ganglion for Acute and Subacute Herpes Zoster Neuralgia: A Randomized Controlled Trial
Brief Title: Esketamine Combined With PRF of DRG for Acute/Subacute Zoster-associated Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Xiaotangshan Hospital (Other); The First Hospital of Fangshan District,Beijing (Other); Beijing Ditan Hospital (Other); Hengshui People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-332-02-04
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster Neuralgia; Esketamine
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine group (Experimental): Esketamine+ PRF group
  Interventions: Drug: esketamine group
- control group (Active Comparator): PRF group
  Interventions: Drug: PRF group

INTERVENTIONS:
Drug: esketamine group — in addition to receiving the combination of PRF of DRG and standardized drug treatment, patients will also undergo a single intravenous infusion of esketamine.
  Other Names: esketamine+PRF+ standardized drug treatment
  Arms: Esketamine group
Drug: PRF group — In the control group, patients will receive PRF+standardized drug treatment. Pulsed radiofrequency (PRF) will be performed on DRG by an designated physician in each participating center. They will be treated with PRF (PMG-230, Baylis Medical Inc.) using a 21-gauge sterilized radiofrequency needle (a 10-cm trocar with a 5-mm active tip, PMF-21-100-5, Baylis Medical Inc.), which are carefully inserted until the needle tip reaches the upper edge of the intervertebral foramen. The parameters of PRF treatment will be set at 42 ℃, 2 Hz with 20 milliseconds current. The standardized drug treatment will include antiviral therapy, anticonvulsant treatment, three-step analgesic therapy
  Other Names: PRF+standardized drug treatment
  Arms: control group

SUMMARY:
To assess the 1-month effects and safety of esketamine - PRF -standardized drug treatment against PRF -standardized drug treatment acute/subacute zoster-associated pain (ZAP) patients.

DETAILED DESCRIPTION:
This study aims to determine whether the addition of esketamine to PRF - standardized drug treatment can improve 1 - month pain control and safety profiles in acute/subacute ZAP patients. The findings may help optimize current treatment strategies for refractory ZAP patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages more than 18 years;
2. Patients with onset of herpes zoster (HZ) rash less than 90 days;
3. HZ affected the spinal nerves (cervical/thoracic/lumbar nerve);
4. Having an average pain score of at least 4 on a Numeric Rating Scale (NRS, 0 = no pain, 10= worst possible pain)；
5. Planned to perform CT-guided PRF treatment of the dorsal root ganglion(DRG).

Exclusion Criteria:

1. Obstructive sleep apnoea syndrome;
2. Those who receive other more invasive treatments, such as radiofrequency thermocoagulation (RFT) of DRG.
3. A history of systemic immune diseases, organ transplantation, or cancers;
4. A history of severe cardiopulmonary, hepatic, renal dysfunction or coagulation function disorder;
5. A history of schizophrenia, epilepsy, or myasthenia gravis, delirium;
6. Comorbid hyperthyroidism or phaeochromocytoma;
7. Recent history of drug abuse;
8. Having contraindications to esketamine;
9. Communication difficulties.
10. Women who are preparing for pregnancy, in the pregnancy or lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
the NRS score at 1 month after treatment. | 1-month period
  The Numeric Rating Scale (NRS) score is a way to quantify the degree of subjective feelings such as pain using numbers. Generally, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain

SECONDARY OUTCOMES:
the NRS score after treatment | at 1 week, 2 weeks, 2 months, 3 months after treatment
  Generally, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain.
the 12-item Short-Form Health Survey (SF-12) score | at 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  Quality of life (QoL) assessed by the SF-12 score (range 0-100, with higher scores indicating better health status)
the Pittsburgh Sleep Quality Index (PSQI) score | at 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  Sleep quality measured by PSQI score (range 0-21, with higher scores indicating poorer sleep quality).
The Patient Global Impression of Change scale (PGIC) | at 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  The proportion of patients with a response of "no change", "minimally improved", "much improved" or "very much improved" on PGIC
Analgesics consumption | at 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  the type of analgesics and analgesics consumption
Safety assessments | at 0 day, 1 day, 1 week, 2 weeks,1 month, 2 months, 3 months
  intraoperative complications, PRF-related complications, esketamine-related complications
success rate | at 1 week, 2 weeks, 1 month, 2 months, 3 months after treatment
  The success rate is defined as more than a 50% reduction in NRS-11 score

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
not yet decided